CLINICAL TRIAL: NCT05441618
Title: Retrospective, Single Center, Single Arm Post Market Clinical Follow-Up (PMCF) Study on the Performance and Safety of Lyoplant® Used for the Replacement and Extension of Connective Tissue Structures in Neurosurgery
Brief Title: Post Market Clinical Follow-Up Study on the Performance and Safety of Lyoplant®
Acronym: LYOPLACE
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2112
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Tumor, Cerebral Ventricle; Tumor, Cerebellar; Aneurysm Cerebral; Trauma, Brain
Keywords: Lyoplant; Retrospective Study; Decompressive Craniectomy; Cerebral Dura Defect; Cerebellar Dura Defect; Spinal Dura Defects
MeSH Terms: conditions — Cerebral Ventricle Neoplasms; Cerebellar Neoplasms; Intracranial Aneurysm; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lyoplant®: Lyoplant® is a pure collagen implant obtained from bovine pericardium. The membrane is used for the replacement and extension of connective tissue structures in neurosurgery.
  Interventions: Device: Lyoplant®

INTERVENTIONS:
Device: Lyoplant® — replacement and extension of connective tissue structures in neurosurgery

SUMMARY:
Retrospective, single center, single arm PMCF study on the performance and safety of Lyoplant® used for the replacement and extension of connective tissue structures in neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Use of investigational device according to Instructions for Use (IfU)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient files from adult patients with indication of surgical diagnosis (e.g. decompressive craniectomy, tumor, aneurysm, trauma etc.) in a single center are revisited and analysed for primary and secondary variables
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Rate of Cerebrospinal Fluid Leakage | at one follow-up ≥ 3 months after surgery
  A Cerebrospinal Fluid (CSF) leakage needs to be confirmed by radiological image evaluation (computed tomography scan, CT or magnetic resonance imaging scan, MRI). It will be documented if the CSF leak was clinically evident or not. A clinically evident CSF leak is defined as clear fluid leaking through the surgical incision or orifice (e.g., rhinorrhea or otorrhea) or as subcutaneous visible and / or palpable fluid accumulation next to or at the site of surgical incision suspected to be CSF. A non-clinically evident CSF leak is defined as CSF accumulation which could be detected only by radiological image evaluation (CT / MRI).

SECONDARY OUTCOMES:
Incidence of re-operations with product relationship | at one follow-up ≥ 3 months after surgery
  e.g. caused by infection, foreign-body-reaction/ hypersensitivity against proteins of bovine origin/ allergic reactions to proteins of bovine origin
Incidence of further (serious) adverse events in chronologic sequence | intra- and postoperative, until follow-up ≥ 3 months after surgery
  Number of further serious adverse events e.g. meningitis, surgical site infection, inflammation rate, hematoma - with focus on events with (possible) relation to the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp E Krauss, Dr., Principal Investigator — Universitätsklinikum Augsburg AöR
Locations (1):
- Universitätsklinikum Augsburg AöR, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No